CLINICAL TRIAL: NCT02757911
Title: A Phase I/II, Non Randomized, Monocentric Open-label Study of Autologous CD34+ Cells Transduced With the G1XCGD Lentiviral Vector in Patients With X-Linked Chronic Granulomatous Disease
Brief Title: Gene Therapy for X-linked Chronic Granulomatous Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G1XCGD.02
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: X-Linked Chronic Granulomatous Disease
Keywords: XCGD
MeSH Terms: conditions — Granulomatous Disease, Chronic

ARMS (1):
- open label (Experimental): X vivo gene therapy
  Interventions: Genetic: X vivo gene therapy

INTERVENTIONS:
Genetic: X vivo gene therapy — Transplantation of patient's autologous CD34+ cells transduced with lentiviral vector containing XCGD gene. The investigational product is patient-specific and corresponds to autologous CD34+ cells transduced ex vivo with the G1XCGD vector. These transduced cells will be cryopreserved until safety testing and infusion into the patient.

SUMMARY:
X-linked chronic granulomatous disease (X-CGD) is a rare genetic disorder, which affects boys. It is a primary immunodeficiency disorder which results from an inability of the white blood cells called phagocytic cells (or phagocytes) to kill invading bacteria and fungi. These cells have difficulty forming the free radicals (most importantly the superoxide radical due to defective phagocyte NADPH oxidase complex) which are important in the killing of ingested pathogens. In X-CGD (which accounts for two thirds of CGD patients), the defect lies in a gene which makes up a critical part of the NADPH-oxidase complex (the catalytic subunit; gp91-phox protein). Therefore they kill bacteria and fungi poorly, and the patients suffer from severe and recurrent infections. This also results in inflammation which can damage parts of the body such as the lung and gut.

In many cases, patients can be adequately protected from infection by constant intake of antibiotics. However, in others, severe life-threatening infections break through. In some cases, inflammation in the bowel or urinary systems results in blockages which cannot be treated with antibiotics, and which may require the use of other drugs such as steroids. Development of curative treatments for CGD is therefore of great importance.

ELIGIBILITY:
Inclusion Criteria:

* Male X-CGD patients >23 months of age. Youngest patients (>1 month and ≤ 23 months) may be enrolled at physician's appreciation; in this case mobilization of peripheral HSC may be replaced by two bone marrow harvests.
* Molecular diagnosis confirmed by DNA sequencing and supported by laboratory evidence for absent or reduction > 70% of the biochemical activity of the NAHPD-oxidase.
* At least one ongoing or resistant or at high risk of relapse severe infection and/or inflammatory complications requiring hospitalisation despite conventional therapy.
* No HLA-matched donor available after 3 months search, unless the risk of waiting for a potential match or for performing an allogeneic transplant is considered unacceptable.
* No co-infection with Human Immunodeficiency Virus (HIV) or hepatitis B virus (HBs Ag positive) or hepatitis C virus (anti-HCV Ab positive).
* Written informed consent for adult patient.
* Parental/guardian and where appropriate child's signed consent/assent.

Exclusion Criteria:

* 10/10 HLA identical (A, B, C, DR, DQ) family or unrelated.
* Contraindication for leukapheresis (anaemia Hb <8g/dl, cardiovascular instability, severe coagulopathy).
* Contraindication for administration of conditioning medication and any component of the Investigational Medicinal Product (IMP) preparation.
* Administration of gamma interferon within 30 days before the infusion of transduced autologous CD34+ cells.
* Participation in another experimental therapeutic protocol within 6 months prior to baseline and during the study period.
* Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful completion of the study.
* Patient/Parent/Guardian unable or unwilling to comply with the protocol requirements.

Min Age: 24 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2034-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the incidence of adverse events | 60 months
Restoration and stability over time of the NADPH functioning granulocytes assessed by a Dihydrorhodamine (DHR) flow cytometry test | 12 months

SECONDARY OUTCOMES:
Clinical improvement | 60 months
  Assessed by: complete physical examination to assess the normalisation of nutritional status, the growth, the development, the decrease in the severity of the infection and/or inflammatory complication at inclusion.
Percentage of transduced CD34+ haematopoietic cells infused and of blood cells over time | 60 months
Immunological reconstitution | 60 months
  Assessed by: evidence of restored neutrophil functionality (DRH test), expression of gp91phox protein by flow cytometry and immunity against bacterial and fungal infections over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane BLANCHE, MD, PHD, Principal Investigator — Hôpital Necker-Enfants Malades
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France